CLINICAL TRIAL: NCT04185116
Title: Improvement in Surgical Performance With 3D High Definition Systems: Olympus VISERA ELITE II 3D
Brief Title: 3D-HD Optic Systems Influence Surgical Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Víctor Turrado-Rodríguez, Gastrointestinal Surgeon, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HCB/2018/1203
Record Dates: First submitted 2019-09-05; First posted 2019-12-04 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Operative Time; Fatigue; Surgery--Complications
Keywords: 3D optic systems; Fatigue; Length of surgery; 3D laparoscopy; Intraoperative complications; Bariatric and metabolic surgery
MeSH Terms: conditions — Fatigue; Intraoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 3D Optic Surgeons (Experimental): Full-trained surgeons randomised into this interventional arm will be performing laparoscopic gastric bypass using a 3D optic system.
  Interventions: Device: 3D Optic System (Olympus VISERA Elite II 3D)
- 2D Optic Surgeons (No Intervention): Full-trained surgeons randomised into this interventional arm will be performing laparoscopic gastric bypass using a 2D optic system.
- 3D Optic Residents (Experimental): 4th and 5th year General Surgery residentes randomised into this interventional arm will be performing laparoscopic gastric bypass using a 3D optic system.
  Interventions: Device: 3D Optic System (Olympus VISERA Elite II 3D)
- 2D Optic Residents (No Intervention): 4th and 5th year General Surgery residentes randomised into this interventional arm will be performing laparoscopic gastric bypass using a 2D optic system.

INTERVENTIONS:
Device: 3D Optic System (Olympus VISERA Elite II 3D) — Use of the 3D Optic System "Olympus VISERA Elite II 3D"
  Arms: 3D Optic Residents; 3D Optic Surgeons

SUMMARY:
Randomized controlled trial in which two different laparoscopic systems: standard 2D and Olympus VISERA Elite II 3D will be compared in terms of laparoscopic skills, length of surgery, intraoperative complications and surgeon's fatigue in a group of senior surgeons and senior residents will be measured when performing laparoscopic Roux-en-Y gastric bypass.

DETAILED DESCRIPTION:
The introduction of minimally invasive surgery has faced the surgeon with some difficulties that were not present in traditional open surgery. The foremost disadvantage of laparoscopy is the loss of depth perception in 2-dimensional (2D) vision while having to operate in a 3-dimensional (3D) space.

Minimally invasive surgery has become the standard approach for most of the abdominal surgical procedures. It is associated with less surgical trauma, faster recovery, shorter hospital stay and better cosmetic results. These advantages have led laparoscopic skills to become a basic competence for general surgery programs. Advanced laparoscopic surgery involves a long learning curve, including demanding minimally invasive skills such as intracorporeal suturing and knot tying.

Video quality is critical for an accurate training. This is especially important for advanced laparoscopic skills training, where high-definition cameras are needed. HD imaging has been shown to provide subjectively improved image for visualization and to improve surgical task performance.

Some authors have investigated the effect of laparoscopic 3-dimensional view, and have demonstrated an improvement in speed, efficiency, optics and handling as well as surgeon's subjective assessment. Moreover, 3D systems have been demonstrated to provide better optical visualization that allows simpler presentation of anatomical structures, which can decrease intraoperative errors and postoperative morbidity secondary to visual distortions and may reduce postoperative fatigue of the surgeon.

The hypothesis of the study is that the length of surgery is reduced with the use of 3D laparoscopic systems compared with 2D laparoscopic systems, the reduction on the length of surgery will be higher on the training surgeons compared with the senior surgeons, and that the use of 3D laparoscopic systems reduces the postoperative fatigue of the surgeons.

In this study a group of full-trained surgeons and of 4th and 5th year General Surgery Residents performing laparoscopic Roux-en-Y Gastric Bypass will be randomized into the use of 2D standard laparoscopic optics or 3D laparoscopic optics.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obesity (BMI > 30)
* Laparoscopic Gastric Bypass candidates

Exclusion Criteria:

* Non-obese patients.
* Candidates to other surgical procedures than laparoscopic gastric bypass

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Duration of Surgery | Day 1
  Total time to perform the jejuno-jejunal anastomosis and closure of the mesenteric defect.

SECONDARY OUTCOMES:
Intraoperative complications | Day 1
  Record of the intraoperative complications that may occur during the procedure (bleeding, bowel injury, mesenteric injury, disruption of the anastomotic suture)
Profile of Mood States (POMS) | Day 1
  Measurement of self-perceived fatigue using the POMS scale
Quick Questionnaire Piper Fatigue Scale (QPFS) | Day 1
  Measurement of self-perceived fatigue using QPFS
Visual Analogue Scale (VAS) - related fatigue | Day 1
  Fatigue measured using the VAS
Postoperative complications | 90 days after surgery
  Classification of the postoperative complications using the Clavien-Dindo Classification

CONTACTS AND LOCATIONS:
Locations (1):
- Victor Turrado-Rodriguez, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gomez-Gomez E, Carrasco-Valiente J, Valero-Rosa J, Campos-Hernandez JP, Anglada-Curado FJ, Carazo-Carazo JL, Font-Ugalde P, Requena-Tapia MJ. Impact of 3D vision on mental workload and laparoscopic performance in inexperienced subjects. Actas Urol Esp. 2015 May;39(4):229-35. doi: 10.1016/j.acuro.2014.09.008. Epub 2014 Nov 12. English, Spanish. PMID 25457567
- [Background] Alaraimi B, El Bakbak W, Sarker S, Makkiyah S, Al-Marzouq A, Goriparthi R, Bouhelal A, Quan V, Patel B. A randomized prospective study comparing acquisition of laparoscopic skills in three-dimensional (3D) vs. two-dimensional (2D) laparoscopy. World J Surg. 2014 Nov;38(11):2746-52. doi: 10.1007/s00268-014-2674-0. PMID 25002241
- [Background] Honeck P, Wendt-Nordahl G, Rassweiler J, Knoll T. Three-dimensional laparoscopic imaging improves surgical performance on standardized ex-vivo laparoscopic tasks. J Endourol. 2012 Aug;26(8):1085-8. doi: 10.1089/end.2011.0670. PMID 22721451
- [Background] Ozsoy M, Kallidonis P, Kyriazis I, Panagopoulos V, Vasilas M, Sakellaropoulos GC, Liatsikos E. Novice surgeons: do they benefit from 3D laparoscopy? Lasers Med Sci. 2015 May;30(4):1325-33. doi: 10.1007/s10103-015-1739-0. Epub 2015 Mar 15. PMID 25772250
- [Background] Curro G, La Malfa G, Caizzone A, Rampulla V, Navarra G. Three-Dimensional (3D) Versus Two-Dimensional (2D) Laparoscopic Bariatric Surgery: a Single-Surgeon Prospective Randomized Comparative Study. Obes Surg. 2015 Nov;25(11):2120-4. doi: 10.1007/s11695-015-1674-y. PMID 25893652
- [Background] Bilgen K, Ustun M, Karakahya M, Isik S, Sengul S, Cetinkunar S, Kucukpinar TH. Comparison of 3D imaging and 2D imaging for performance time of laparoscopic cholecystectomy. Surg Laparosc Endosc Percutan Tech. 2013 Apr;23(2):180-3. doi: 10.1097/SLE.0b013e3182827e17. PMID 23579515
- [Background] Andrade E, Arce C, Torrado J, Garrido J, De Francisco C, Arce I. Factor structure and invariance of the POMS Mood State Questionnaire in Spanish. Span J Psychol. 2010 May;13(1):444-52. doi: 10.1017/s1138741600003991. PMID 20480710
- [Background] Cuesta-Vargas AI, Fernandez-Lao C, Cantarero-Villanueva I, Castro-Sanchez AM, Fernandez-de-Las Penas C, Polley MJ, Arroyo-Morales M. Psychometric properties of the QuickPIPER: a shortened version of the PIPER Fatigue scale. Eur J Cancer Care (Engl). 2013 Mar;22(2):245-52. doi: 10.1111/ecc.12022. Epub 2013 Jan 16. PMID 23320955